CLINICAL TRIAL: NCT01325766
Title: Yoga as a Therapy for Adolescents and Young Adults With Cystic Fibrosis: A Pilot Study
Brief Title: Study of Yoga as a Therapy for Cystic Fibrosis (CF) Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seattle Children's Hospital (Other)
Collaborators: Firland Foundation (Unknown)
Responsible Party: Jennifer Ruddy MD, Seattle Children's Hospital, University of Washington Medical Center
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13424
Record Dates: First submitted 2011-03-16; First posted 2011-03-30 (Estimated); Last update posted 2011-03-30 (Estimated); Status verified 2011-03

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Yoga
MeSH Terms: conditions — Cystic Fibrosis | interventions — Yoga

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Yoga (immediate start) group (Active Comparator): This arm will start yoga sessions immediately after screening and will continue sessions for 8 weeks. This group will then continue with home yoga for an additional 8 weeks.
  Interventions: Other: Yoga
- Yoga (waitlist) group (Active Comparator): This arm will continue regular CF therapies for 8 weeks and will start yoga sessions at week 9.
  Interventions: Other: Yoga

INTERVENTIONS:
Other: Yoga — Yoga 2 sessions per week for 8 weeks

SUMMARY:
Cystic fibrosis (CF) is a lung disease that affects 30,000 children and adults in the US. Incorporation of regular exercise into the lives of patients with CF is of interest because it may improve lung function and quality of life. Yoga is an activity that may benefit patients with CF in many ways including strengthening muscles of breathing, improving lung function, and reducing stress which could improve quality of life and adherence to therapies. Yoga has been shown to be beneficial in patients with other lung diseases such as asthma, but has not yet been studied in CF.

The investigators hypothesize that yoga will be an activity that is safe and tolerable for CF patients 12 to 25 years of age. The primary aim is to investigate the safety and tolerability of an 8 week yoga program for patients with CF. The secondary aim is to determine the effect of yoga on many aspects of CF disease including respiratory symptoms, adherence to regular CF therapies, quality of life, lung function, exercise tolerance, and nutritional status.

The long-term goal is to use the data obtained in this study to design a future study of the efficacy of yoga in a larger population of CF patients at multiple CF centers. This research has the potential to influence the prevention and treatment of CF by providing data which could be used to help understand the most appropriate and beneficial type of physical activity for CF patients.

ELIGIBILITY:
Inclusion Criteria:

o Diagnosis of CF by: Sweat chloride ≥60meq/L on two occasions or CFTR genotype with two CF disease-causing mutations and one or more phenotypic features of CF

* Age ≥12 and ≤25 years
* FEV1 ≥40 % predicted at screening visit
* Informed consent and assent

Exclusion Criteria:

* Wheezing on auscultation of the chest at the enrollment visit
* Oxygen saturation < 90 % at the enrollment visit
* Initiation of treatment with oral, inhaled or intravenous antibiotics for an acute respiratory infection in the 2 weeks preceding the enrollment visit
* Pregnancy
* History of lung transplant
* Practiced yoga regularly (≥1 time per week) in the month prior to enrollment
* Current enrollment in a therapeutic clinical trial
* Condition or situation which, in the opinion of the investigator, would affect the ability of the patient or family to complete study procedures

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-10 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety | 16 weeks
  Determine if a yoga program is safe for CF patients by monitoring for adverse events throughout the study.
Pain Scores on the Visual Analog Scale as a measure of tolerability | 16 weeks
  Participants will be given a tolerance questionnaire after each yoga session which will assess their degree of musculoskeletal and chest pain on a visual analog scale. Vital signs will also be measured before and after each yoga session.

SECONDARY OUTCOMES:
Quality of Life | 16 weeks
  This will be assessed with the Cystic fibrosis quality of life questionnaire-revised. This is a CF specific quality of life outcome measure and will be administered at each study visit.
Respiratory symptoms | 16 weeks
  This will be assessed using a cystic fibrosis respiratory symptom diary that will taken once per week at home throughout the study.
Treatment adherence | 16 weeks
  This will be assessed by participants taking a treatment adherence questionnaire once per week at home. Questions are asked regarding compliance with other CF therapies.
Pulmonary function | 16 weeks
  Pulmonary function will be monitored by spirometry at the screening visit and at both study visits. Participants will be assessed for response to bronchodilator at the screening visit. If there is a positive response, post-bronchodilator testing will be done again at the last study visit.
Ease of breathing | 16 weeks
  This will be assessed by the ease of breathing score which is a measure of shortness of breath after activity. This will be done at screening and at each study visit.
BMI | 16 weeks
  BMI will be assessed at each study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Ruddy, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States